CLINICAL TRIAL: NCT02143206
Title: Modifying Exercise for the COPD Patient With Arthritic Limitations to Improve Compliance in a Pulmonary Rehab Program
Brief Title: Modifying Exercise for the COPD Patient
Status: Completed | Type: Observational
Sponsor: Angela N Fellner PhD CCRP (Other)
Responsible Party: Sponsor-Investigator, Angela N Fellner PhD CCRP, Clinical Research Specialist, TriHealth Inc.
Organization: TriHealth Inc. (Other)
Other Study IDs: 12026-12-024
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Arthritis; Pain
Keywords: Chronic Obstructive Pulmonary Disease; Pain; Arthritis; Dyspnea; Exercise; Aerobic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Arthritis; Pain; Dyspnea; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Exercise Method: Patients attend exercise 80 minute exercise sessions of which 30 minutes includes aerobic exercise on a NuStep and Biodex elliptical machine. Patients pain levels are scored when using the NuStep then when using the Biodex and these scores are compared to determine which machine give the best outcome for pain management

SUMMARY:
This study will test whether using the Biodex BioStep Semi Recumbent Elliptical for the chronic obstructive pulmonary disease (COPD) patient with arthritic limitations will improve participation in a pulmonary rehab program compared to the Nustep elliptical. The main outcome of participation will be measured by the number of exercise sessions the patient is able to complete during their pulmonary rehabilitation program. In addition, distance walked in six minutes, dyspnea score, rate of perceived exertion (RPE) score, Pain Scale Index score, and finally, the Dartmouth Quality of Life index (DQL) will be assessed in both groups. It is believed that the new machine will provide better overall outcomes compared to the traditional machine.

DETAILED DESCRIPTION:
A Prospective cohort study of 25 COPD patients with osteoarthritis undergoing an exercise plan in a pulmonary rehab program. Patient pain level, clinical outcomes, and ultimately, quality of life outcomes will be assessed in order to assess whether future compliance for COPD arthritic patients will occur in an exercise rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* COPD Patient
* Osteoarthritic limitations in upper or lower extremities, or spine
* Forced Expiratory Volume (FEV)1 less than 70%
* Forced Expiratory Volume/Forced Vital Capacity (FEV/FVC) ratio less than 70%

Exclusion Criteria:

* Patients with rheumatoid arthritis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 25 COPD patients (total N = 50) with osteoarthritis undergoing an exercise plan in a pulmonary rehab program.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of Exercise Sessions Attended | 2 years

SECONDARY OUTCOMES:
Distance Walked | 6 minutes

OTHER OUTCOMES:
Dyspnea Score | Two years
Rate of Perceived Exertion | 30 minutes
Pain Index Score | 30 minutes
Dartmouth Quality of Life Index | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Craig Eisentrout, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth Fitness and Health Pavilion, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No